CLINICAL TRIAL: NCT01838070
Title: Regulatory Post-Marketing Surveillance (PMS) Study for AVAXIM 160U (Hepatitis A Vaccine)
Brief Title: Regulatory Post-Marketing Surveillance Study for Hepatitis A Vaccine (AVAXIM 160U)
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: HAF85; U1111-1127-7211 (Other: WHO)
Record Dates: First submitted 2013-04-18; First posted 2013-04-23 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Hepatitis A
Keywords: Hepatitis A; Hepatitis A vaccine; AVAXIM 160U
MeSH Terms: conditions — Hepatitis A; Hepatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: Participants that has received AVAXIM 160U vaccine administered under the routine practice according to Summary of Product Characteristics

SUMMARY:
This safety surveillance study is being conducted in accordance with Korea Food and Drug Administration (KFDA) "Basic standard for reexamination of new drug".

Primary objective:

* To assess the safety of AVAXIM 160U (Hepatitis A vaccine) administered under the routine practice, according to Korea Food and Drug Administration "Basic standard for reexamination of new drug" based on the pharmaceutical law in Korea.

DETAILED DESCRIPTION:
The study will be conducted under the real clinical practices in accordance with Korea Food and Drug Administration "Basic standard for reexamination of new drug".

No vaccine will be provided and/or administered as part of this protocol, however only participants that has received AVAXIM 160U vaccine administered under the routine practice according to Summary of Product Characteristics will be part of the surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 16 years and older
* Informed consent signed by the subject and by parent or legal representative for subject aged 16 to 19 years
* Informed consent sign by subject for subject aged of 20 year of age and older
* Receipt of AVAXIM 160U according to Summary of Product Characteristics (SmPC).

Exclusion Criteria:

* Contraindications to vaccination according to AVAXIM 160U Summary of Product Characteristics (SmPC)
* Subject is known to be pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche or post-menopausal for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence for at least 4 weeks prior to the vaccination until at least 4 weeks after)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received AVAXIM 160U (Hepatitis A Vaccine) according to Summary of Product Characteristics (SmPC)
Sampling Method: Non-Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2013-04; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety profile in terms of solicited and unsolicited adverse events following the administration of AVAXIM 160U vaccine | Day 0 up to 30 Days post-vaccination
  Solicited injection site: Pain, Erythema, and Swelling: Solicited Systemic Reactions: Fever (temperature), headache, and myalgia. Unsolicited averse events including non serious and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur SA
Locations (1):
- Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Oh Y, Thollot Y, Bravo C. Post-Marketing Surveillance of Hepatitis A Virus Vaccine (Avaxim(R) 160U) in South Korea from 2011 to 2015. Infect Dis Ther. 2019 Mar;8(1):105-112. doi: 10.1007/s40121-019-0230-9. Epub 2019 Jan 23. PMID 30673992
- See also: Related Info — http://www.sanofipasteur.com